CLINICAL TRIAL: NCT03437213
Title: The Immunomodulatory Effect of Bilateral Paravertebral Block and Total Intravenous Anesthesia in Spine Surgery.
Brief Title: The Immune Modulation of Bilateral Paravertebral Block and Propofol in Spine Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alaa Mazy Mazy (Other)
Responsible Party: Sponsor-Investigator, Alaa Mazy Mazy, associate professor of anesthesia and surgical intensive care, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MD/17.12.52
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Immune Suppression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total intravenous anesthesia group (Experimental): propofol, and fentanyl-based regimen.
  Interventions: Drug: Total intravenous anesthesia group
- Total intravenous plus block group (Active Comparator): ultrasound guided paravertebral block before induction then propofol and fentanyl maintenance.
  Interventions: Drug: Total intravenous plus block group

INTERVENTIONS:
Drug: Total intravenous anesthesia group — Induction of general anesthesia with fentanyl, (1mcg / kg), propofol (1-2 mg / kg), atracurium (0.5 mg / kg), intubation. Anesthesia maintained using Propofol (4-6) mg/kg/h, fentanyl (0.5-1) μg/kg/h. to be modified according to analgesic needs and hemodynamics. 10mg atracurium when the 2nd twitch of train of four appears.
  Arms: Total intravenous anesthesia group
Drug: Total intravenous plus block group — Ultrasound guidance identifies the paravertebral space using a linear high-frequency (10-12 MHz) probe in the transverse plane in the midline, rotate the probe to the longitudinal plane, and scan in a medial-to-lateral direction. Locate the desired segment shift from the cephalad aspect of the sacrum. The transverse scan will show a hyperechoic outline of the vertebral spinous and transverse processes. Use the loss of resistance technique. Bilaterally inject (5ml) bupivacaine 0.5% for each segment. Induction of anesthesia after 30 minutes with fentanyl, (1mcg / kg), propofol (1-2 mg / kg), atracurium (0.5 mg / kg),then prone position.
  Arms: Total intravenous plus block group

SUMMARY:
General anesthesia has an important effect on inflammatory cytokines. Inhalational agents as isoflurane and sevoflurane attenuate immune function expressed by neutrophil chemoattractant-1 as well as inflammatory enzyme and also they reduce inflammatory cascade. Total intravenous anesthesia (TIVA) based on using propofol suppresses the inflammatory response caused by surgery to a greater extent because Propofol affects the balance between pro-inflammatory and anti-inflammatory cytokines, increasing production of the anti-inflammatory cytokine IL-10 and at the same time reducing the increase of IL-6 during the perioperative period. It also alters expression of nitric oxide and inhibits neutrophil function. TIVA has many advantages such as; fewer side effects, earlier discharge, better patient satisfaction, faster recovery, less nausea and vomiting and reduced muscle relaxant requirements. Paravertebral block has an important role in the inflammatory and immune response. The paravertebral block can decrease perioperative inflammation and prevent immune suppression. Also, it can attenuate the cytokine response and reduce acute stress response caused by surgery. Decrease inflammation processes, improve surgery result, limit the duration of hospital stay, decrease post-operative fatigue and reduce postoperative complications.

DETAILED DESCRIPTION:
Spine surgery is characterized by an elevation in levels of the inflammatory cytokines such as interleukin IL-6, IL-1β, and IL-17. These cytokines promote chemokine production and changes in cell phenotype which lead to activation of T and B cells, macrophages, neutrophils, and mast cells further amplifying the inflammatory cascade. Different analgesic modalities are used for pain management during and after spine surgery as narcotic analgesics, nonsteroidal anti-inflammatory drugs, Paracetamol and neuraxial techniques like intrathecal drug administration, epidural analgesia and paravertebral block. In this study, Paravertebral Block is used as a new and recent analgesic strategy for spine surgery. It has the advantage of higher success rate and analgesic efficacy, less risk of neurological complications than most other regional anesthetic techniques, less nausea, vomiting, and constipation compared with opioid-based analgesic techniques, urinary retention does not occur, unlike neuraxial techniques and intense block of both the sympathetic and somatic nerves. This study will be conducted with the hypothesis that the addition of paravertebral block as an analgesic regimen with total intravenous anesthesia (propofol-based) will have a better Immunomodulatory effect in patients undergoing posterior lumbar spine fixation surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for primary fixation of posterior lumbar spine surgery.
* American Society of Anesthesia statuses I or II patients.
* Single or double level lumbar spine fixation.
* Fixed surgical team.

Exclusion Criteria:

1. Patient refusal or uncooperative Patient.
2. History of allergy to any anesthetic agents will be used in the study.
3. Local sepsis.
4. Abnormal coagulation test results.
5. Usage of antiplatelet therapy.
6. Demyelinated neurological diseases as multiple sclerosis.
7. Mental retardation, psychotropic drug consumption.
8. Recurrent spine fixation.
9. Severe coronary or peripheral artery disease.
10. Severe cardiac disease, renal or hepatic failure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-25 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Serum levels of interleukin 6 (IL-6). | 24 hours postoperative
  picogram/milliliter using ELISA techniques. Measured Basal: 30 minutes before starting anesthesia, 2 hours after starting surgery, 8 and 24 hours from the end of surgery postoperative.
Serum levels of interleukin 1β (IL-1β). | 24 hours postoperative.
  picogram/milliliter using ELISA techniques. Measured Basal: 30 minutes before starting anesthesia, 2 hours after starting surgery, 8 and 24 hours from the end of surgery postoperative.

SECONDARY OUTCOMES:
Total leukocyte count. | 24 hours postoperative.
  Number multiplied by 1000 /micro liter, measured Basal: 30 minutes before starting anesthesia, 2 hours after starting surgery, 8 and 24 hours from the end of surgery postoperative.
Absolute neutrophil count. | 24 hours postoperative.
  Number multiplied by 1000 /micro liter, measured Basal: 30 minutes before starting anesthesia, 2 hours after starting surgery, 8 and 24 hours from the end of surgery postoperative.
Neutrophil-Lymphocyte-Ratio (N/L ratio). | 24 hours postoperative.
  ratio. Measured Basal: 30 minutes before starting anesthesia, 2 hours after starting surgery, 8 and 24 hours from the end of surgery postoperative.
Serum cortisol level. | 24 hours postoperative.
  Micro-gram per deciliter by immunoassays techniques. Measured Basal: 30 minutes before starting anesthesia, 2 hours after starting surgery, 8 and 24 hours from the end of surgery postoperative.
C-reactive protein serum level. | Basal: 30 minutes before starting anesthesia, 2 hours after starting surgery, 8 and 24 hours from the end of surgery postoperative.
  milligram per liter using ELISA techniques.
the time to the first analgesic request. | 24 hours postoperative.
  hours.
Total morphine consumption. | 24 hours postoperative.
  milligram.
The total amount of blood loss. | Intraoperative; from the start of anesthesia to the end of surgery (minutes).
  milliliter, estimated by weighing the swabs and blood suction loss.
The amount of allogenic blood transfusion. | Intraoperative; from the start of anesthesia to the end of surgery (minutes).
  Unites.
the duration of surgery. | intraoperative.
  Minutes, from the start of anesthesia to the extubation time.
The length of hospital stay. | 1-5 days postoperative.
  Days, Starts from 0 hour postoperative time until patient discharge from the hospital.
Mean arterial pressure | Basal 30 minutes preoperative, 5 minutes after intubation, 5 minutes after prone position, after 30, 60, 90, 120, 150, 180 min intraoperative. Postoperative, at 6, 12, 24 h after operation.
  millimeter mercury
Heart rate | Basal 30 minutes preoperative, 5 minutes after intubation, 5 minutes after prone position, after 30, 60, 90, 120, 150, 180 min intraoperative. Postoperative, at 6, 12, 24 h after operation.
  Beats per minute.
Numeric Pain Scale | 24 hours postoperative.
  A scale from 0 to 10, where 0= no pain, and 10= worst imaginable pain. The patient describe subjective pain feeling in a number from (0- 10). Measured basal 30 minutes before anesthesia, 30 min after para-vertebral block. postoperative at 6, 12, 24 hours. then after 1st, 2nd, 3rd months postoperative.
The European Quality of Life-5 Dimensions measures. | After 1st, 2nd, 3rd months postoperative.
  The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: 1, no problems, 2, slight problems, 3, moderate problems, 4, severe problems, and 5, extreme problems. by ticking a box. the final result is a 5 number code that represents the health state.
Basal Metabolic Rate | After 1st, 2nd, 3rd months postoperative.
  Calories. by the Mifflin - St Jeor equation equals = 10 × weight (kg) + 6.25 × height (cm) - 5 × age(y) + 5
The rate of postoperative complications | Postoperative within 72 hours after surgery.
  the percent of the complications: thromboembolic events, surgical complications (Wound infection, bleeding, wound hematoma and neurological complication), postoperative fever, and nausea with vomiting.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided